CLINICAL TRIAL: NCT03204981
Title: Intramural Needle Ablation for the Treatment of Refractory Ventricular Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 17-1899
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Ventricular Arrythmia
Keywords: intramural needle ablation; ventricular arrhythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intramural Needle Ablation (Experimental)
  Interventions: Device: Intramural Needle Ablation; Procedure: Ablation

INTERVENTIONS:
Device: Intramural Needle Ablation — The needle-tipped ablation catheter that will be used for the IN ablation uses radiofrequency like a standard RF ablation catheter, but delivers energy through an extendable/retractable needle.
Procedure: Ablation — standard ablation

SUMMARY:
This study will examine the safety and efficacy of intramural needle ablation (INA) in the treatment of intramural ventricular arrhythmias in patients for whom standard RF ablation has been unsuccessful. The clinical team hypothesize that the increased current density and improved rates of transmural lesion creation seen with intramural needle ablation will lead to successful arrhythmia termination with minimal or no increased risk of complication.

DETAILED DESCRIPTION:
Radiofrequency (RF) ablation is the most commonly employed method for the catheter treatment of cardiac arrhythmias. Myocardial scar serves as the most frequent substrate for the genesis of both atrial and ventricular arrhythmias. Such scar frequently contains surviving myocyte bundles interspersed with fibrotic tissue, which leads to slow conduction. Areas of denser fibrosis cause conduction block. When appropriately arranged, conduction through or around these scars leads to the creation of a "reentry" circuit through which an arrhythmia is generated and maintained. Each reentry circuit contains within it an area called the isthmus, a portion of the circuit located in a position intimately related to the scar border zone. Electrical activation travels slowly through the isthmus before breaking out into normal myocardium. Ablation at the site of an isthmus will terminate a reentrant tachycardia.

A variety of techniques, including electroanatomic mapping and activation, entrainment, and substrate mapping, are employed during electrophysiologic (EP) study to identify areas of myocardial scar and potential isthmus sites. Points or lines of ablation using RF energy are then created in an attempt to interrupt the reentry circuit. Typically, RF energy is applied via a catheter tip electrode to the endocardial or epicardial surface of the heart and grounded via an electrode pad placed on the patient's skin. RF energy in this setting is dispersed through the entirety of the tissue between catheter tip and grounding pad. The standard 7-French, 4-mm tip catheters are highly successful at ablating circuits located within a few millimeters of the catheter tip. A focal, 1mm area of resistive heating occurs within the myocardium immediately in contact with the catheter tip; myocardial cell death occurs several millimeters more deeply through passive, conductive heating, which spreads outward from the contact point.

While the standard catheter is effective at the ablation of superficial arrhythmias, it has proven more problematic when used for deep myocardial sites or for creating transmural lesions. A number of alternatives have been developed in an attempt to access these sites. 8-mm or 10-mm catheter tips are able to create larger zones of resistive heating, delivering direct RF energy to a larger area of myocardium. A larger interface between catheter tip and blood improves cooling and allows for the delivery of more power without a rise in impedance.The clinical use of these larger catheters can, however, be limited by rapid temperature rises at the catheter-tissue interface, resulting in thrombus formation, char, and "steam pop" rupture of the endocardial surface. The use of irrigated ablation catheters have improved upon the ability to deliver RF energy without a sustained rise in impedance. Both open irrigated- and closed-loop irrigated catheters circulate saline along the catheter tip-myocardial interface, allowing for continued delivery of RF current without thrombus formation at the endocardial surface. Intramyocardial temperature rises accordingly without a concomitant endocardial temperature surge, creating larger and deeper myocardial ablation zones. Transcoronary ethanol ablation has also been employed with moderate success in patients with arrhythmias resistant to endocardial catheter ablation.This technology, however, grants only limited control over the size of the resulting infarct and is restricted by the need for perfusion of the scar zone by an accessible coronary artery.

Nevertheless, there remain occasions in which an arrhythmia cannot be eliminated by standard ablation techniques. This is seen most frequently due to deep intramural ventricular tachycardia, sometimes encountered following myocardial infarction. Both standard and alternative ablation strategies are frequently either unavailable or inadequate for termination of these arrhythmias.

Initial experience with an electrically active needle electrode have demonstrated that radiofrequency ablative energy can effectively create lesions of homogeneous necrosis. Needle electrodes have been used experimentally from the epicardial surface, from the endocardium ex vivo and in vivo in an internally irrigated form. It has been shown that the use of a narrow-gauge non-irrigated endocardial needle ablation catheter creates very narrow but deep lesions due to the small electrode size. Catheters featuring a retractable needle tipped electrode with intramyocardial saline infusion have also shown promise as a means of accessing deep myocardial circuits in ventricular tachycardia ablation.18

The proposed study will further examine the role of INA in patients with ventricular arrhythmias resistant to standard ablation techniques.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with any of the following criteria: a) monomorphic ventricular tachycardia (VT); b) frequent ventricular arrhythmia (defined as unifocal PVCs, couplets, non-sustained VT) with a PVC burden ≥13%, or is causing a decline in left ventricular (LV) ejection fraction to <40%; or c) previous failed ablation for one or more of the criteria above.
* ≥ 15 years of age.
* Left ventricular (LV) ejection fraction > 10% as estimated by echocardiography, contrast ventriculography or radionuclide imaging within the past 90 days.
* Clinical indication for catheter ablation of VT
* Intramural ventricular arrhythmias not terminable with standard ablation once enrolled in the Intramural Needle Ablation study or previous failed ablation within 6 months prior to enrollment.
* Ability to understand the requirements of the study and sign the informed consent form.
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements.
* Projected lifespan greater than 1 year.

Exclusion Criteria:

* History of MI or CABG within 6 weeks.
* NYHA Class IV CHF.
* Patients with idiopathic ventricular arrhythmias defined as VT or PVCs that occur without evidence of structural heart disease and that are not causing significant depression of LV function.
* Women known to be pregnant or to have positive beta-HCG.
* Definite protruding left ventricular thrombus on pre-ablation echocardiography or other imaging modalities.
* Contraindication to heparin
* Allergy to radiographic contrast dye.
* Unstable angina that is not due to frequent or incessant VT.
* Acute non-cardiovascular illness or systemic infection.
* Thrombocytopenia (platelet count < 50,000 mm3) or coagulopathy.
* Cardiogenic shock unless it is due to incessant VT.
* Unable to sign consent.
* Projected lifespan of < 1 year.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tedrow UB, Kurata M, Kawamura I, Batnyam U, Dukkipati S, Nakamura T, Tanigawa S, Fuji A, Richardson TD, Kanagasundram AN, Koruth JS, John RM, Hasegawa K, Abdelwahab A, Sapp J, Reddy VY, Stevenson WG. Worldwide Experience With an Irrigated Needle Catheter for Ablation of Refractory Ventricular Arrhythmias: Final Report. JACC Clin Electrophysiol. 2023 Aug;9(8 Pt 2):1475-1486. doi: 10.1016/j.jacep.2023.05.014. Epub 2023 May 19. PMID 37278684
- [Derived] Dukkipati SR, Nakamura T, Nakajima I, Oates C, Narui R, Tanigawa S, Sljapic T, Whang W, Koruth JS, Choudry S, Schaeffer B, Fujii A, Tedrow UB, Sapp JL, Stevenson WG, Reddy VY. Intramural Needle Ablation for Refractory Premature Ventricular Contractions. Circ Arrhythm Electrophysiol. 2022 May;15(5):e010020. doi: 10.1161/CIRCEP.121.010020. Epub 2022 Apr 27. PMID 35476455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intramural Needle Ablation
Started | 52
Completed | 46
Not Completed | 6
Not completed — Physician Decision | 2
Not completed — Screen failures (no inducible VT or PVCs) | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.26 (16.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 41
  More than one race | 0
  Unknown or Not Reported | 6
Patients with Ventricular Tachycardia (VT) [Count of Participants; unit: Participants] | 24
Patients with Premature Ventricular Contractions (PVCS) [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Freedom From Ventricular Arrhythmia at 6 Months
Description: Number of participants with VT and number of participants with PVCs who had freedom from ventricular arrhythmia at 6 months for participants who had ablation performed using the experimental Needle ablation catheter versus standard ablation catheter.
  Needle - patient had ablation performed using the experimental Needle ablation catheter.
  Registry - patient had ablation using a standard ablation catheter and did not need additional ablation using the Needle catheter.
Time Frame: 6 months
Population: participants analyzed for those with VT and those with PVCs
Measure: Count of Participants; unit: Participants
Groups:
- Participants With VT: Participants with Ventricular Tachycardia (VT)
- Participants With PVCs: Participants with Premature Ventricular Contractions (PVCS)
Arm/Group | Participants With VT | Participants With PVCs
Number analyzed (Participants) | 24 | 22
Participants
  Needle: number analyzed (Participants) | 13 | 16
  Needle | 8 | 4
  Registry: number analyzed (Participants) | 11 | 6
  Registry | 5 | 2

2. Secondary Outcome: Number of Events of Procedural Complications
Description: Number of events of procedural complications
Time Frame: at 6 months
Population: There were 21 participants that experienced a procedural complication event.
Measure: Number; unit: events
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 21
events | 29

3. Secondary Outcome: Number of Participants With Post-ablation Inducibility
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 46
Participants | 2

4. Secondary Outcome: Time to Termination
Time Frame: Day 1
Population: The researchers were only able to capture data on termination times for six patients. Many number of patients did not have termination. Others had termination, but the study team was not able to ascertain the time to termination.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 6
seconds | 322.16 (189.91)

5. Secondary Outcome: Total Duration of Intramural Needle Ablation
Description: Total duration of intramural needle ablation for patient who had ablation performed using the experimental Needle ablation catheter.
Time Frame: Day 1
Population: Data analyzed for participants who had experimental needle ablation.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 29
minutes | 47.14 (40.51)

6. Secondary Outcome: Total Number of Intramural Needle Ablations
Description: Total Number of Intramural Needle Ablations for patient had ablation performed using the experimental Needle ablation catheter.
Time Frame: Day 1
Population: Data analyzed for participants who had experimental needle ablation.
Measure: Mean (Standard Deviation); unit: ablations
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 29
ablations | 11.2 (9.0)

7. Secondary Outcome: All-cause Mortality
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intramural Needle Ablation
Number analyzed (Participants) | 46
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intramural Needle Ablation
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 15/52
Other Adverse Events (participants affected / at risk) | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intramural Needle Ablation (N=52)
Acute respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Acute Stroke (Nervous system disorders) | 1
Chest pain with recurrent VT (Cardiac disorders) | 1
CHF (Cardiac disorders) | 3
Complete Heart Block (Cardiac disorders) | 1
Hypervolemia with right ventricular failure and increased right sided pressures (Cardiac disorders) | 1
Hypotension (General disorders) | 1
LAA thrombus (Cardiac disorders) | 1
Metabolic encephalopathy with hyperammonemia (Nervous system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericardial effusion with hypotension (Cardiac disorders) | 1
Repeated falls (General disorders) | 1
Right Femoral artery dissection (Vascular disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vasovagal syncope (General disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intramural Needle Ablation (N=52)
Apical thrombus (Cardiac disorders) | 1
Bleed from groin site (Vascular disorders) | 1
Cardiac Sarcoidosis (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Complete Heart Block (Cardiac disorders) | 1
Fever (Infections and infestations) | 1
Gastrointestinal bleed (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hematuria with UTI and urinary retention (Renal and urinary disorders) | 1
Hypotension (General disorders) | 2
Left bundle branch block (Cardiac disorders) | 1
Left femoral artery dissection (Vascular disorders) | 1
Left groin hematoma (Vascular disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Orthostatic hypotension with lightheadedness and tremors (General disorders) | 1
Paraphimosis (Renal and urinary disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Renal failure (Renal and urinary disorders) | 1
UTI (Renal and urinary disorders) | 1
Ventricular tachycardia with intermittent chest pain and dyspnea (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03204981/Prot_SAP_000.pdf